CLINICAL TRIAL: NCT05418517
Title: The Incidence of Hospital Acquired Pneumonia in Patients Who Undergo Temporary Tracheostomy With Oromaxillofacial Resection and Reconstruction for Head and Neck Cancer.
Brief Title: Hospital Acquired Pneumonia in Temporary Tracheostomy
Acronym: HAP
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: King's College London (Other)
Responsible Party: Principal Investigator, Rachel Wijayarathna, Highly specialist physiotherapist - head & neck oncology, Guy's and St Thomas' NHS Foundation Trust
Other Study IDs: IRAS ID295395
Record Dates: First submitted 2022-06-10; First posted 2022-06-14 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Head and Neck Cancer; Tracheostomy Complication; Hospital-acquired Pneumonia; Surgery
MeSH Terms: conditions — Head and Neck Neoplasms; Healthcare-Associated Pneumonia | interventions — Tracheostomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- oromaxillofacial surgery: Patients who underwent oromaxillofacial surgery
  Interventions: Procedure: Tracheostomy; Procedure: Overnight intubation

INTERVENTIONS:
Procedure: Tracheostomy — temporary tracheostomy insertion
Procedure: Overnight intubation — Patient who had overnight intubation

SUMMARY:
Medical condition or disease under investigation:

Oromaxillofacial surgery in head and neck cancer

Purpose of research:

Retrospective data analysis identifying hospital acquired pneumonia in patients who undergo temporary tracheostomy with oromaxillofacial surgery and free flap reconstruction

Primary objective:

Undertake an adequately powered, robustly designed observational cohort study that describes the rates of hospital acquired pneumonia in patients who undergo a tracheostomy and those that undergo overnight intubation during oromaxillofacial surgery for HNC.

Secondary objective:

To investigate whether smoking history, respiratory history (COPD, asthma) or size of tumour are associated with an increased risk of developing hospital acquired pneumonia.

Number of Subjects/Patients: 193 Study Type: Observational cohort

Main Inclusion Criteria:

Patients who underwent oromaxillofacial resection with free flap reconstruction and tracheostomy from 1st January 2018 to 31st December 2018.

Patients who underwent oromaxillofacial resection with free flap reconstruction and with overnight intubation from 1st January 2014 to 31st December 2014

Statistical Methodology and Analysis:

A power calculation has been used to determine the sample size required for statistical analysis of data. Statistical significance for rates of HAP will be tested between the two groups.

DETAILED DESCRIPTION:
Trial objectives and purpose

* To select patients according to a pre-defined set of inclusion and exclusion criteria
* Collect pre-determined quantitative data relevant to the study question using hospital medical records
* Describe patient demographic data and explore any relationship between these and the development of a HAP
* Asses rates of HAP using historical medical data and pre-defined criteria that identifies hospital acquired pneumonia
* Describe rates of HAP in patients who did not have a tracheostomy inserted for maxillofacial surgery with free flap reconstruction
* Describe rates of HAP in patients who did have a tracheostomy inserted for maxillofacial surgery with free flap reconstruction

Study Design In 2017, a new maxillofacial surgeon was appointed to Guy's & St Thomas' NHS Foundation Trust who's preference was to insert a temporary tracheostomy for all patients undergoing oromaxillofacial surgery with free flap reconstruction. Prior to this there was a wide variation in case selection with the majority of patients undergoing overnight intubation. Since subsequent practice has now changed and all patients now undergo tracheostomy insertion within OMFS, a prospective design is not possible, therefore, a single site retrospective observational design will be adopted, allowing data from two cohorts of patients identified to be collected within a feasbile timeframe dictated by the module deadlines. Electronic and paper notes of patients from cohorts before and after the change in maxillofacial surgical practice (2014 and 2018) will be screened.

ELIGIBILITY:
Subject inclusion criteria

* Patients who underwent maxillofacial resection with free flap reconstruction and tracheostomy from 1st January 2018 to 31st December 2018.
* Patients who underwent maxillofacial resection with free flap reconstruction and with endotracheal intubation from 1st January 2014 to 31st December 2014
* Patients over the age of 18

Subject exclusion criteria

* Patients who did not undergo maxillofacial resection with free flap reconstruction and tracheostomy from 1st January 2018 to 31st December 2018 - not relevant and will not answer the study question
* Patients who did not undergo maxillofacial resection with free flap reconstruction and with endotracheal intubation from 1st January 2014 to 31st December 2014 - not relevant and will not answer the study question
* Patients under the age of 18

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient who have head and neck cancer and require oromaxillofacial resection and reconstruction with a free flap
Sampling Method: Non-Probability Sample
Enrollment: 193 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Hospital acquired pneumonia | 7 days post surgery
  Development of hospital acquired pneumonia according to BMJ best practice 'hospital acquired pneumonia' (non covid-19) diagnosis criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Guy's and St Thomas' NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No plan to share data

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-24): https://cdn.clinicaltrials.gov/large-docs/17/NCT05418517/Prot_SAP_000.pdf